CLINICAL TRIAL: NCT06248983
Title: Transmission Of Respiratory Tract microOrganisms In a School Environment - the TORTOISE-study
Brief Title: Transmission Of Respiratory Tract microOrganisms In a School Environment
Acronym: TORTOISE
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Principal Investigator, Simon P Jochems, PhD, Associate professor, Leiden University Medical Center
Other Study IDs: P23.094; NL85480.058.23 (Registry Identifier: CCMO - toetsingonline.nl)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Tract Infections; Transmission; Microbial Colonization; Viral Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal epithelial lining fluid will be sampled using a nasosorption device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Observational study, therefore no intervention that is administered.

SUMMARY:
Through contact with peers in daycare and (primary)school young children play a large role in spreading respiratory pathogens. In this study the investigators will investigate this transmission, the subsequent colonization and infection dynamics, and their association with clinical symptoms and local immune response through dense minimally-invasive sampling. This study will allow us a unique insight into the transmission-, infection-, and colonization-potential of the respiratory pathogens.

DETAILED DESCRIPTION:
Respiratory tract infections impose a large burden of disease upon the world. Pneumonia remains the leading infectious cause of death in children under five worldwide. Known causative agents of pneumonia include, but are not limited to, Spn, Haemophilus influenzae (HI), Moraxella catarrhalis (MC) and viruses such as the Respiratory Syncytial Virus (RSV) and the influenza virus. These microorganisms are regularly found in the upper respiratory tract (URT) without causing severe disease. Colonization of the URT is thought to be important both for immune boosting and to provide competition for other potential harmful colonizers.

This study aims to provide insights into the processes and key host immune and microbiota factors that determine the infection kinetics, transmission and development of immunity during such infections. Furthermore, this study will enable us to closely study the transmission of commonly found microorganisms in an environment that is prone to transmission, the close quarters of school classes in which young children and their teachers spend a large part of their time.

Research within this specific population (risk-group and high transmitting group), young children and their teachers, is warranted. This is due to differences in the pediatric and adult mucosal immune system and infection and transmission dynamics, while animal models not being directly translatable to the human situation.

In this study the investigators will perform dense, longitudinal sampling within groups of closely interacting children and their teachers to study spread and colonization. Furthermore, by determining a range of biomarkers along with profiling the respiratory microbiome the investigators can look for markers predicting colonization and symptomatic infection.

By measuring airobiome through the EDC and air samples collected by a pollensniffer the investigators can measure local exposure to environmental microbes, human pathogens and pollen. This will allow us to compare immune responses and correlate this with clinical symptoms of RTI.

ELIGIBILITY:
There are 2 sets of eligibility criteria, one for participating children and one for participation teachers.

Children:

Inclusion Criteria:

* Within age-limit
* attending primary school

Exclusion Criteria:

* Insufficient proficiency of their parents in Dutch or English language

Teachers:

Inclusion Criteria:

* Adult teacher of participating primary school class

Exclusion Criteria:

* Insufficient proficiency in Dutch or English language

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children attending primary school, age 4-7 (year 1-2 of primary education) and their teachers. The investigators aim to include minimal 80% of children in a given class. In total the investigators aim to include three classes within one season.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Classroom transmission- and colonization-rate of Streptococcus pneumoniae in young children. | 8 weeks
  To answer the primary objective the investigators will record pneumococcus carriage over time at a serotype level using qPCR. This will lead to a categorical variable with the following levels for each included serotype, per participant: never infected (no Spn detected during the sampling period), already colonized (Spn detected at the start of the sampling period), new colonization (Spn not detected at the start of the sampling period, but detected in the course of the sampling period) or re-colonization (same Spn serotype detected during sampling period with at least 3 samples in between not detecting Spn).
  A transmission event will be defined as a Spn serotype that is observed in at least one child in the class and at a later timepoint also observed in one or more other children, as long as this is within 1 week of it being present in first child.

SECONDARY OUTCOMES:
Transmission and colonization rates of other URT pathogens in a classroom setting. | 8 weeks
  Presence, transmission and/or introduction of common URT commensals/pathogens will be recorded and lead to categorical variables similar to the primary study parameter. Subtyping/sequencing will be performed where deemed relevant (rhinovirus, influenza virus etc.) to elude the source to the extent possible.
Nasal immune response in response to exposure, infection or colonization by URT microbes. | 8 weeks
  Local host immune response in response to colonization/infection of URT by pathogens and potential differences in response between different pathogens will be measured using tools as ELISA or multiplex technologies, such as Olink and Luminex. The investigators will focus on innate and adaptive inflammatory markers. The investigators will also measure antibodies against pathogens using tools as ELISA and antigen arrays.
The relationship between clinical symptoms of RTI's, host immune responses, microbiome and URT pathogens. | 8 weeks
  Clinical symptoms of RTI's will be recorded in categorical variables (yes/no).The microbiome will be measured by RNA sequencing. Microbial products will be measured by tools like mass spectrometry.
pollen and bacterial presence (airobiome) in classroom environment via electrostatic dust fall collector and pollensniffer to differentiate between RTI and hay fever. | 8 weeks
  Pollen (counts and species) and microbial presence in classroom environment will be measured via Electrostatic Dust Collector and active air sampling using a pollensniffer.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Leiden University Medical Centre, Leiden, Zuid-Hollend

IPD SHARING:
Plan to Share IPD: No